CLINICAL TRIAL: NCT06748430
Title: Assessment of the Effect of Different Varieties of Grapes on Postprandial Glycemia and Insulinemia
Brief Title: Effects on Glycemia and Insulinemia of Different Grape Varieties
Acronym: SUGARGAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Principal Investigator, Santiago Navas, Researcher at the Center for Nutrition Research, Universidad de Navarra, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SUGARGAP
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Healthy; Glycaemic Response Measurements
Keywords: Grape variety; Glycaemic response; metabolome; insulin response

STUDY DESIGN:
Intervention Model Description: The group of subjects will go through the three visits of the study in the same order. All subjects will consume the same variety at the same time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Variety 1 (timpson) (Placebo Comparator): Reference variety
  Interventions: Other: Grape variety control
- Variety 2 (18INV-1438-10) (Active Comparator): First comparator
  Interventions: Other: Grape variety 1
- Variety 3 (18-1465-110) (Active Comparator): Second comparator
  Interventions: Other: Grape variety 2

INTERVENTIONS:
Other: Grape variety control — Reference grape variety
  Arms: Variety 1 (timpson)
Other: Grape variety 1 — First grape variety to evaluate
  Arms: Variety 2 (18INV-1438-10)
Other: Grape variety 2 — Second grape variety to evaluate
  Arms: Variety 3 (18-1465-110)

SUMMARY:
The goal of this intervention study is to examine the glucose increase in blood, during 2 hours after consuming different varieties of grapes, in men and women with normal or excess body weight. The main question it aims to answer is:

can a variety of red grape reduce the glucose curve compared to a reference variety?

Participants will have to attend the Center for nutrition research facilities in three occasions, fasted for at least 8 hours. Once there, they will be measured and monitored. A canula will be inserted and once they finish eating 300g of grapes, blood extractions will be performed at minutes 15, 30, 60, 90 and 120.

DETAILED DESCRIPTION:
The main purpose of this study is to evaluate how the glucose and insulin curves develop after consuming different grapes varieties. Still, we also want to evaluate how the serum metabolome changes with the three varieties after 120 minutes. Therefore, a metabolomic study will be done in samples of volunteers at this time point.

The intervention is longitudinal and in three arms (one per variety). Due to the harvest of the different varieties, it cannot be crossover, but each subject will consume the three varieties.

At each visit, the subjects will undergo the same schedule:

* Arrival in a fasting state of at least 8 hours.
* Insertion of cannula and extraction of fasting samples
* Consumption of approximately 300 g of grapes (50 g of Carbohydrates).
* Extraction of blood samples at 15, 30, 60, 90 and 120 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Baseline glycaemia between 70 and 100 mg/dL
* BMI between 18.5 kg/m2 and 29.9 kg/m2.
* Absence of disease or alterations related to gastrointestinal status.
* Signed written informed consent.

Exclusion Criteria:

* Glycaemic levels out of the reference inclusion criteria (below 70 or over 100 mg/dL)
* Subjects presenting BMI out of the limits set.
* Subjects with unstable body weight the three months prior the start of the study (+/- 3 Kg)
* Subjects not able to attend the preestablished visits
* Women pregnant or lactating
* Subjects undergoing pharmacological treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Glycaemic response | 0 minutes
  Assessment of serum glucose evolution after consuming 50 g of carbohydrates in grapes
Glycaemic response | 15 minutes
  Assessment of serum glucose evolution after consuming 50 g of carbohydrates in grapes
Glycaemic response | 30 minutes
  Assessment of serum glucose evolution after consuming 50 g of carbohydrates in grapes
Glycaemic response | 60 minutes
  Assessment of serum glucose evolution after consuming 50 g of carbohydrates in grapes
Glycaemic response | 90 minutes
  Assessment of serum glucose evolution after consuming 50 g of carbohydrates in grapes
Glycaemic response | 120 minutes
  Assessment of serum glucose evolution after consuming 50 g of carbohydrates in grapes
Insulinemic response | 0 minutes
  Assessment of serum insulin evolution after consuming 50 g of carbohydrates in grapes
Insulinemic response | 15 minutes
  Assessment of serum insulin evolution after consuming 50 g of carbohydrates in grapes
Insulinemic response | 30 minutes
  Assessment of serum insulin evolution after consuming 50 g of carbohydrates in grapes
Insulinemic response | 60 minutes
  Assessment of serum insulin evolution after consuming 50 g of carbohydrates in grapes
Insulinemic response | 90 minutes
  Assessment of serum insulin evolution after consuming 50 g of carbohydrates in grapes
Insulinemic response | 120 minutes
  Assessment of serum insulin evolution after consuming 50 g of carbohydrates in grapes
Insulin Resistance Index (HOMA-IR) response | 0 minutes
  Assessment of insulin resistance evolution after consuming 50 g of carbohydrates in grapes
Insulin Resistance Index (HOMA-IR) response | 15 minutes
  Assessment of insulin resistance evolution after consuming 50 g of carbohydrates in grapes
Insulin Resistance Index (HOMA-IR) response | 30 minutes
  Assessment of insulin resistance evolution after consuming 50 g of carbohydrates in grapes
Insulin Resistance Index (HOMA-IR) response | 60 minutes
  Assessment of insulin resistance evolution after consuming 50 g of carbohydrates in grapes
Insulin Resistance Index (HOMA-IR) response | 90 minutes
  Assessment of insulin resistance evolution after consuming 50 g of carbohydrates in grapes
Insulin Resistance Index (HOMA-IR) response | 120 minutes
  Assessment of insulin resistance evolution after consuming 50 g of carbohydrates in grapes
Metabolome composition | 120 minutes
  Metabolomic analysis after grapes consumption

SECONDARY OUTCOMES:
Total cholesterol | 0 minutes
  Serum total cholesterol in fasting state
LDL - cholesterol | 0 minutes
  Serum LDL-cholesterol in fasting state
HDL-cholesterol | 0 minutes
  Serum HDL-cholesterol in fasting state
Triglycerides | 0 minutes
  Serum triglycerides in the fasting state
ALT | 0 minutes
  Serum ALT levels in fasting state
AST | 0 minutes
  Serum AST levels in fasting state

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Navas-Carretero, PhD, Principal Investigator — University of Navarra
Locations (1):
- Center for Nutrition Research. University of Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Undecided